CLINICAL TRIAL: NCT04031729
Title: Aspirin in Adults With Nonalcoholic Fatty Liver Disease
Brief Title: Aspirin for the Treatment of Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tracey G. Simon, MD, Instructor in Medicine and Gastroenterology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P001809
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis
Keywords: Aspirin; Liver Disease; Anti-inflammatory
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin (Experimental): Low-dose (81mg) aspirin tablets
  Interventions: Drug: Aspirin 81 mg
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81mg tablets will be given once daily, for the duration of the clinical trial.
  Arms: Aspirin
Drug: Placebo oral tablet — Identical, blinded placebo tablets will be given once daily, for the duration of the clinical trial.
  Arms: Placebo

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD), defined by fatty infiltration of the liver in the absence of excess alcohol consumption, affects an estimated 30% of adults in the United States. A proportion of people with NAFLD will develop progressive, inflammatory nonalcoholic steatohepatitis (NASH), which can progress to liver cirrhosis and liver failure. NAFLD is expected to be the most common indication for liver transplantation by the year 2020. We hypothesize that among adults with NAFLD, aspirin will reduce intrahepatic lipid content, as quantified by 1H magnetic resonance spectroscopy (1H-MRS).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 70 years
* NAFLD, defined by confirmed hepatic steatosis by imaging or by liver biopsy, in the absence of other causes of hepatic steatosis or significant alcohol consumption. If liver imaging or biopsy has not been performed clinically, liver ultrasound assessment will be performed as part of the screening visit.
* Early-stage liver fibrosis, defined as fibrosis less than or equal to Fibrosis Stage 3 (F3), confirmed by either (1) a recent liver biopsy or (2) a recent elastography / Fibroscan study. If no recent biopsy or elastography/Fibroscan have been performed, a Fibroscan will be performed as part of the screening visit.

Exclusion Criteria:

* Liver fibrosis stage > 3
* Current aspirin use
* Contraindications to aspirin use
* Contraindications to magnetic resonance imaging (MRI)
* Pregnancy or desire to become pregnant
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey G Simon, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simon TG, Wilechansky RM, Stoyanova S, Grossman A, Dichtel LE, Lauer GM, Miller KK, Hoshida Y, Corey KE, Loomba R, Chung RT, Chan AT. Aspirin for Metabolic Dysfunction-Associated Steatotic Liver Disease Without Cirrhosis: A Randomized Clinical Trial. JAMA. 2024 Mar 19;331(11):920-929. doi: 10.1001/jama.2024.1215. PMID 38502074

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 40 | 40
Completed | 37 | 34
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 36 | 73
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 46.6 [24 to 70] | 49.3 [25 to 70] | 47.9 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Black or African American, non-Hispanic | 1 | 0 | 1
  Hispanic or Latino | 6 | 6 | 12
  White, non-Hispanic | 30 | 33 | 63
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Baseline hepatic lipid content (%) by 1H_MRS [Mean (Standard Deviation); unit: percentage of hepatic lipid content] | 39.1 (26.1) | 31.4 (24.8) | 35.0 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Intrahepatic Lipid Content, by 1H-MRS
Description: Absolute percentage change in intrahepatic lipid content, quantified by 1H-MRS
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Mean absolute percentage change
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 40 | 40
Mean absolute percentage change | -6.6 [-11.9 to -1.3] | 3.6 [-1.7 to 8.9]

2. Secondary Outcome: Relative Change in Intrahepatic Lipid Content
Description: Relative percentage point change in intrahepatic lipid content
Time Frame: 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Mean percentage point change
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 40 | 40
Mean percentage point change | -8.8 [-28.3 to 10.8] | 30.0 [10.4 to 49.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each trial participant from the date of screening to the final 6-month study visit date.
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/40
Other Adverse Events (participants affected / at risk) | 12/40 | 12/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=40) | Placebo (N=40)
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=40) | Placebo (N=40)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Arthralgias (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Other infection (Infections and infestations) | 1 (1) | 1 (1)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Atherosclerosis (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT04031729/Prot_SAP_000.pdf